CLINICAL TRIAL: NCT04503889
Title: The Effect of Transauricular Electrical Vagal Nerve Stimulation on Temporal Summation of Heat Pain in Patients With Chronic Low-back Pain
Brief Title: The Effect of Transauricular Electrical Vagal Nerve Stimulation on Temporal Summation of Pain in Patients With Back Pain
Acronym: TVNS_TSP_LBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: BB 095/16
Record Dates: First submitted 2020-07-31; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Pain Intensity
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessor will be unaware regarding the type (real or sham) taVNS intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real taVNS intervention (Experimental): taVNS will be administered to cymba conchae of both ears using ECO2-TENS device
  Interventions: Device: Transauricular electrical vagal nerve stimulation; Device: taVNS sham
- Sham (Sham Comparator): aVNS will be administered to lobes of both ears using ECO2-TENS device
  Interventions: Device: Transauricular electrical vagal nerve stimulation; Device: taVNS sham

INTERVENTIONS:
Device: Transauricular electrical vagal nerve stimulation — transauricular electrical vagal nerve stimulation will be applied to the cymba conchae of both ears using ECO2 TENS device (manufactured by Schwa-Medico GmbH/Germany) with currency intensity of max 10 mA and current frequency 2/100 Hz.
Device: taVNS sham — ECO2 TENS device (manufactured by Schwa-Medico GmbH/Germany)

SUMMARY:
The effect of transauricular electrical vagal nerve stimulation (taVNS) will be studied on temporal summation of heat pain (TSP) in 30 patients with chronic low-back pain and in 30 heathy volunteers. Participants will receive either taVNS or sham stimulation before and during TSP induction in a randomized crossover manner. The participants will be unaware regarding the type of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic low-back pain
* age 30-60 yrs old
* without heart disease
* low-back pain intensity at least 4 out of 10 points measured using NRS-10
* without cognitive deficits (Mini Mental State Shake < 23)

Exclusion Criteria:

* opioid medication
* more than 1 low-back surgery
* sensory of motor neurological deficits at the level of back pain
* spinal stenosis
* diabetic polyneuropathy
* skin pathology at the site (cymba conchae) of stimulation

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-23 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Unpleasantness of pain | Continuously 5 minutes during the experimental heat pain stimulation
  Perceived unpleasantness of pain, which participants will rate continuously during the repetitive heat stimulation using a computerized visual analogue scale (CoVAS, Medoc Advanced Medical Systems, Ramat Yishai, Israel) ranging from 0 (= not unpleasant at all) to 100 (= intolerable pain)

SECONDARY OUTCOMES:
Heart rate | 10 minutes (before, during and after stimulation of heat pain)
  Heart rate (bpm)
blood pressure | 10 minutes (before, during and after stimulation of heat pain)
  non-invasive measurement of systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Taras Usichenko, MD, PhD, Study Chair — University Medicine of Greifswald
Locations (1):
- University Medicine of Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: Undecided